CLINICAL TRIAL: NCT00388804
Title: Randomized Trial of External Beam Radiation With or Without Short-Course Hormonal Therapy in Intermediate Risk Prostate Cancer Patients
Brief Title: External Beam Radiation Therapy (EBRT) With or Without Hormonal Therapy in Prostate Cancer
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Slow accrual.
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2003-0819
Record Dates: First submitted 2006-10-15; First posted 2006-10-17 (Estimated); Results first posted 2012-08-08 (Estimated); Last update posted 2012-08-08 (Estimated); Status verified 2012-06

CONDITIONS: Prostate Cancer
Keywords: Prostate Cancer; External Beam Radiotherapy; Radiation Therapy; Hormone Therapy; Bicalutamide; Casodex; Leuprolide; Lupron; Goserelin; Zoladex; Flutamide; EBRT
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Radiotherapy; bicalutamide; Leuprolide; Goserelin; Flutamide; Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- RT Group 1 (Active Comparator): Radiation Therapy (RT) over 8 1/2 weeks: 42 treatments, 5 days per week with 2 days rest in between.
  Interventions: Procedure: Radiation Therapy; Behavioral: Questionnaire
- RT Group 2 + Hormone Therapy (Active Comparator): Radiation Therapy over 8 1/2 weeks; + Hormone Therapy (Bicalutamide 50 mg orally/day or Flutamide 250 mg orally 3 times daily on first 21-30 Days) + Leuprolide (22.5 mg Intramuscularly (IM)/every 3 months or 7.5 mg IM monthly) or Goserelin (10.8 mg subcutaneously every 3 months or 3.6 mg subcutaneously monthly)
  Interventions: Procedure: Radiation Therapy; Drug: Bicalutamide; Drug: Leuprolide; Drug: Goserelin; Drug: Flutamide; Behavioral: Questionnaire

INTERVENTIONS:
Procedure: Radiation Therapy — Radiation treatment given over about 8 1/2 weeks; 42 treatments, 5 days per week with 2 days rest in between.
  Other Names: RT; XRT
Drug: Bicalutamide — 50 mg By Mouth (PO) Daily
  Other Names: Casodex
  Arms: RT Group 2 + Hormone Therapy
Drug: Leuprolide — 22.5 mg Intramuscularly (IM) Every 3 Months or 7.5 mg IM Every 1 Month
  Other Names: Lupron
  Arms: RT Group 2 + Hormone Therapy
Drug: Goserelin — 10.8 mg Subcutaneously Every 3 Months or 3.6 mg Subcutaneously Every 1 Month
  Other Names: Zoladex
  Arms: RT Group 2 + Hormone Therapy
Drug: Flutamide — 250 mg by mouth three times daily on first 21-30 Days. May be used instead of Bicalutamide.
  Arms: RT Group 2 + Hormone Therapy
Behavioral: Questionnaire — Questionnaires regarding health-related quality of life given before therapy begins, each taking about 15 minutes to complete.
  Other Names: Survey

SUMMARY:
Primary Objective:

* To assess the possible improvement in prostate specific antigen (PSA) outcome of short course androgen suppression therapy in conjunction with dose-escalation intensity modulated radiation therapy (IMRT), 3D conformal radiation therapy (3D-CRT), or proton therapy over IMRT, 3D-CRT, or proton therapy alone in prostate cancer patients traditionally considered at intermediate risk for PSA failure following conventional local therapy. PSA failure will be the primary endpoint.

Secondary Objectives:

* To assess local control, freedom from distant metastasis, and overall survival.
* To study the impact of radiation therapy and/or hormone therapy on health-related quality of life measures using the Expanded Prostate Cancer Index Composite-Short Form 12-American Urological Association Symptom Index (EPIC-SF12-AUASI: http://roadrunner.cancer.med.umich.edu/epic/).
* To assess prognostic value of pretreatment serum testosterone as well as the decrease in hemoglobin from neoadjuvant hormone therapy.
* To assess prognostic value of pretreatment biomarkers on subsequent post-treatment clinical outcomes.

DETAILED DESCRIPTION:
Prior patient studies have shown that short-term hormone therapy (about 4 months) before and during radiation therapy can benefit patients with bulky tumors or locally-advanced prostate tumors. These prior results have been used to justify a potential benefit for using short-term hormone therapy combined with radiation therapy for patients with less bulky or less advanced prostate cancers. However, the combination of hormone therapy and radiation has not been shown to definitively benefit patients with your level of prostate cancer. Furthermore, these older studies used relatively low doses of radiation by today's standards, and hormone therapy may be of no benefit when using higher doses of radiation. Researchers want to study the use of combination hormone therapy and radiation therapy in the treatment of your level of prostate cancer.

If you are eligible to take part in this study, you will be randomly assigned (as in the toss of a coin) to one of 2 treatment groups. There is an equal chance of being assigned to either treatment group.

If you are assigned to Group 1, you will receive high-dose radiation treatment given over about 8 1/2 weeks. During this period, you will receive up to 42 treatments, 5 days per week with 2 days rest in between. There will be no treatment on weekends. This is the current standard schedule of treatment for prostate cancer patients. A radiation treatment planning session will be done before the actual radiation treatments. This planning session will be used to get images of your prostate and other pelvic organs to help plan the radiation fields. The planning session involves a computed tomography (CT) scan that takes about 40-45 minutes. During this time, about 3 special, permanent tattoo marks will be placed on your skin using ink. The tattoo marks will help with daily setup and positioning of the radiation fields. These marks are small and about the size of a freckle.

If you are assigned to Group 2, you will receive the same radiation therapy as participants in Group 1, but you will also receive hormone therapy with bicalutamide (Casodex) and either leuprolide (Lupron) or goserelin (Zoladex). The hormone therapy includes a total of 2 injections or shots (leuprolide or goserelin) given every 3 months and a pill (bicalutamide) that is taken once per day for the first 21 to 30 days. Flutamide, which is taken three times per day for the first 21-30 days, may be used instead of bicalutamide. The choice of hormone therapy will be left up to your treating physician. You will receive hormone therapy for a full 6 months. Hormonal treatment will begin about 2 months before radiation therapy is due to start and continue for 2 months during radiation therapy, with the last phase of hormone treatment for 2 months after radiation therapy.

No matter which group you are assigned to, you will be given questionnaires to study health-related quality of life. These questionnaires will take about 15 minutes to complete and will be given to you before therapy begins. Within 1-2 weeks before starting radiation therapy, you will answer a health-related quality of life questionnaire (Expanded Prostate Cancer Index Composite-SF12-AUASI). Participants who are receiving hormonal therapy will also be given this questionnaire within one week before hormonal therapy. During radiotherapy, you will be examined every week, and severe side effects and reactions will be recorded using the modified acute toxicity scale. During radiotherapy, you also will be given the EPIC-26 Short Form at Weeks 4 and 8.

After you finish radiation therapy, you will be given the EPIC-SF12-AUASI every 3 months for the first year, every 6 months for the next 2 years, and then once a year after that. This may be done in person, by phone or by mail.

Prostate specific antigen (PSA) and testosterone levels will be checked before therapy begins. These blood tests will require about 1 teaspoon of blood. They will be checked before radiation therapy begins, but will not be checked during your radiation treatment. Your PSA and testosterone levels will be rechecked at 3 to 6 month intervals after the radiation therapy is done for the first 2 years. PSA will be checked every 6 months for the Years 3 and 4, and once a year for Year 5.

If you have worsening of disease or have intolerable side effects, you may elect to remove yourself from the prescribed treatment, but you may still be followed as part of the study.

You will be asked to return for follow-up testing in the form of physical exam every 6 months for the first 2 years and once each year after that. The purpose of the follow-up visits and tests is to check the response of your cancer to treatment. If the PSA or physical exam shows that the disease has not gone away completely or has come back, you may have repeat staging with a bone scan, pelvic CT or magnetic resonance imaging (MRI), and repeat prostate biopsy.

You will be watched for the condition of your disease for at least 4-5 years with follow-up visits and PSA tests. If you are willing to return for follow-up visits beyond 5 years, then you will continue to receive long term follow-up and be observed and advised about your illness, according to your individual needs.

ELIGIBILITY:
Inclusion Criteria:

1. Biopsy proven prostate cancer within last 12 months. Pathology must be reviewed at M.D. Anderson Cancer Center (MDACC).
2. 1992 American Joint Committee on Cancer (AJCC) clinical stage T1c-2b on digital rectal exam with biopsy Gleason sum of 7 and Prostate-Specific Antigen (PSA) < 20 ng/mL (i.e. PSA 19.99 ng/mL or less)
3. 1992 AJCC clinical stage T2b on physical exam with biopsy Gleason sum of 7 or less and/or PSA < 20 ng/ml
4. 1992 AJCC clinical stage T1c-2b on digital rectal exam with biopsy Gleason sum of 7 or less and PSA > 10 but less than 20 ng/ml (i.e. 10.01-19.99 ng/mL). PSA used for protocol eligibility should be obtained within 30 days of protocol enrollment.
5. No evidence of metastatic disease on bone scan within 3 months of study enrollment.
6. No evidence of metastatic disease on pelvic computed tomography (CT) or magnetic resonance imaging (MRI) within 3 months of study enrollment.
7. Zubrod performance status < 2.
8. Must be able to understand protocol and adhere to follow-up initially at 3 months post-radiation and then at 6 month intervals for first two years and annually thereafter.
9. Patient must be able to undergo adequate daily trans-abdominal ultrasound localization (B.A.T.) or other image-guided localization of the prostate during radiation course.
10. Patients will be allowed to participate in other protocols if they are eligible and the other protocols do not interfere with participation in this protocol.

Exclusion Criteria:

1. Patients who do not meet the inclusion criteria. Specifically, patients with all the following features: clinical T1c-2a and Gleason sum of 6 and PSA </= 10 ng/ml. Patients with one or more of the following features: clinical T2c, or Gleason 8-10, or PSA > 20 ng/ml are not eligible.
2. Prior androgen suppression therapy. (Prior finasteride and saw palmetto allowed but must be discontinued prior to enrollment. Biopsy and PSA must be documented prior to finasteride use.)
3. Previous or concurrent malignancies other than basal or squamous cell skin cancers unless disease-free for 5 years or more.
4. Prior pelvic radiation or chemotherapy. Patients who received chemotherapy for non-prostate cancer malignancies over 5 years prior will be eligible.
5. Prior or planned radical prostate surgery.
6. Patients with clinical evidence or biopsy-proven extracapsular extension, seminal vesicle involvement, or lymph node involvement will be excluded. Patients with radiographic evidence of nodal or bone metastasis will be excluded.
7. Other histologies such as small cell carcinoma, sarcomatoid or ductal variants are not eligible.
8. Patients with any Gleason grade 5 disease on biopsy will not be eligible.

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2005-02; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew K. Lee, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- UT MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: UT MD Anderson Cancer Center — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment period: 02/16/2005 to 09/08/2010. All recruitment was at UT MD Anderson Cancer Center.
Pre-assignment Details: Of the 39 enrolled participants, one participant was excluded from the trial before assignment to groups.
Period: Overall Study
Arm/Group | RT Group 1 | RT Group 2 + Hormone Therapy
Started | 17 | 21
Completed | 17 | 21
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | RT Group 1 | RT Group 2 + Hormone Therapy | Total
Number analyzed (Participants) | 17 | 21 | 38
Age Continuous [Median (Full Range); unit: years] | 66.3 [53 to 78] | 64.5 [48 to 73] | 65.3 [48 to 78]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 17 | 21 | 38
Region of Enrollment [Number; unit: participants]
  United States | 17 | 21 | 38

OUTCOME MEASURES:

1. Primary Outcome: Prostate Specific Antigen (PSA) Failures
Description: Baseline + Post-radiation PSA levels at three month intervals for initial two years then every 6 months thereafter. Participants with a rising PSA and no evidence of local or distant recurrence considered PSA failures.
Time Frame: 3 months up to 2 years
Population: One person was not treated and therefore excluded from the analysis.
Measure: Number; unit: participants
Arm/Group | RT Group 1 | RT Group 2 + Hormone Therapy
Number analyzed (Participants) | 17 | 21
participants | 0 | 0

ADVERSE EVENTS:
Time Frame: 4 years and 9 months
Arm/Group | RT Group 1 | RT Group 2 + Hormone Therapy
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/21
Other Adverse Events (participants affected / at risk) | 4/17 | 1/21
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | RT Group 1 (N=17) | RT Group 2 + Hormone Therapy (N=21)
Urinary frequency (Renal and urinary disorders) | 2 | 1 — 2 of 17 (11.8%) in Arm 1 experienced urinary frequency 1 of 21 (4.7% in Arm 2 experienced urinary frequency
Urinary incontinence (Renal and urinary disorders) | 1 | 0 (0)
Dysuria (Renal and urinary disorders) | 1 | 0
Diarrhea (Gastrointestinal disorders) | 1 | 0
Alanine transaminase (ALT) (Metabolism and nutrition disorders) | 1 | 0 — Grade I elevated ALT, no relationship to protocol treatment
Aspartate transaminase (AST) (Metabolism and nutrition disorders) | 1 | 0 — Grade I elevated AST, possibly related to protocol treatment

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No